CLINICAL TRIAL: NCT06022315
Title: Role of Gastrointestinal Appetite Hormones in the Success of Body Mass Loss Interventions Based on Exercise Combined With Calorie-restricted Diets With Different Fat and Carbohydrate Content
Brief Title: Impact of Macronutrient Composition of Energy-restricted Diet and Exercise on Body Composition and Appetite Hormones.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer Human Nutrition School of Medicine, Dentistry and Nursing College of Medical, Veterinary & Life Sciences University of Glasgow, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Glasgow
Record Dates: First submitted 2023-07-30; First posted 2023-09-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Gastrointestinal Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- restricted high carbohydrate low fat diet with exercise training program (Experimental): exercise training combined with the consumption of caloric restricted high CHO-low FAT diet. The interventions will last for four weeks.
  Interventions: Combination Product: caloric restrction high carbohydrate low fat diet with exercise training program
- restricted High fat low carbohydrate diet with exercise training program (Experimental): exercise training with consumption of caloric restricted low CHO-high FAT diet. The interventions will last for four weeks.
  Interventions: Combination Product: caloric restrction high fat low carbohydrate diet with exercise training program

INTERVENTIONS:
Combination Product: caloric restrction high carbohydrate low fat diet with exercise training program — Subjects will perform 3 sessions/week of brisk walking for four weeks at a heart rate corresponding to 85-90% of the lactate threshold. The duration of exercise sessions will increase from 30 minutes to 45 minutes in week 2 and from 45 minutes to 60 minutes in weeks 3 and 4.
  Experimental diets will be calorie-restricted and provide 70% of estimated daily energy requirements. In the high CHO-low FAT diet, carbohydrates, fat, and protein will provide 60%, 25%, and 15% of individually predicted daily energy intake, respectively. Variety (n=7) of daily menus for calorie-restricted high FAT-low CHO diet will be provided and menus for high CHO-low FAT diet on pasta, rice, oats, fruit, and vegetable.During the intervention, participants will be encouraged to avoid alcohol consumption and only the maximum amount of two units will be allowed per week.
  Arms: restricted high carbohydrate low fat diet with exercise training program
Combination Product: caloric restrction high fat low carbohydrate diet with exercise training program — Subjects will perform 3 sessions/week of brisk walking for four weeks at a heart rate corresponding to 85-90% of the lactate threshold.The duration of exercise sessions will increase from 30 minutes to 45 minutes in week 2 and from 45 minutes to 60 minutes in weeks 3 and 4.
  Experimental diets will be calorie-restricted and provide 70% of estimated daily energy requirements. In the low CHO-high FAT diet, the proportion of energy provided by CHO, fat, and protein will consist of 25%, 60%, and 15%, respectively. Variety (n=7) of daily menus for calorie-restricted low CHO-high FAT diet will be provided and menus for high FAT-low CHO group will be based on meat, fish, cheese, butter, and nuts.During the intervention, participants will be encouraged to avoid alcohol consumption and only the maximum amount of two units will be allowed per week.
  Arms: restricted High fat low carbohydrate diet with exercise training program

SUMMARY:
The main aim of this study is to investigate the effect of energy-restricted low and high-carbohydrate diet combined with exercise training on appetite regulatory hormones, subjective appetite and energy intake in overweight and obese women. In addition, since the macronutrient composition of meals and exercise impacts biomarkers of cardiovascular disease, the impact of these interactions on metabolic risk factors of cardiovascular diseases will also be investigated .

DETAILED DESCRIPTION:
This will be a block randomised parallel study, with one group of participants undergoing exercise training combined with the consumption of a calorie-restricted high CHO-low FAT diet and another group undergoing exercise training with consumption of a calorie-restricted low CHO-high FAT diet. The interventions will last for 4 weeks. Prior to and after the interventions participants will undergo a 5-hour experimental trial, which will involve body composition measurements by the D2O method, appetite hormones, insulin via blood collection and subjective appetite via a visual analogue scale. During the experimental trials, participants will consume breakfast and ad libitum buffet-style lunch.

Prior to the first experimental trial, participants will be subjected to a screening process followed by a preliminary exercise test in the metabolic research unit at New Lister Building (NLB), Glasgow Royal infirmary (GRI). Participants will also be asked to record their food and drink consumed for 4 days (3 weekdays and 1 weekend) prior to and during the four last days of the intervention. By following this step, individual diets will be designed based on participants preferences with restricted energy intake and different macronutrient compositions. Dietary intake records will allow a comparison of participants' calorie intake before and after the intervention.

During intervention participants will consume either energy-restricted low CHO-high FAT or energy-restricted high CHO-Low FAT diet and exercise (brisk walking) while wearing a heart rate monitor 3 times a week after 5 minutes of warm-up, and 5 minutes The duration of the brisk walking will increase after week one from 30 to 45 minutes and to 60 minutes at week three and four. Participants will be advised to cool down after the brisk walking session. During the intervention, participants will be encouraged to avoid alcohol consumption. In case this was not possible, a maximum amount of two units will be allowed per week.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female
* BMI of ≥25.0 kg/m2.
* stable body weight for at least three months preceding the study

Exclusion Criteria:

* smokers and have
* irregular menstruation cycle,
* use any type of medication,
* exercising more than 75min a week,
* are pregnant or lactating.
* on any dietary supplements at the time of the study,
* are vegetarian or are following any diet other than the typical Western diet.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal appetite hormones | 240 minutes through study completion
  Plasma concentration (pg/ml) before and after intervention during experimental trials

SECONDARY OUTCOMES:
Total body water | at baseline and after 3 hours
  Saliva sample (ml) before and after 3 hours of drinking D2O water during experimental trials
subjective appetite | 240 minutes through study completion
  Assess via visual analogue scale (100mm)
energy intake | 3 days before and after intervention
  Energy intake (Kcal) during intervention
Insulin | 240 minutes through study completion
  Plasma concentration (mU/L)before and after intervention during experimental trials

CONTACTS AND LOCATIONS:
Overall Officials: Taibah Almesbehi, Principal Investigator — University of Glasgow, New lister Building, Glasgow, Scotland, United kingdom, G31 2ER
Locations (1):
- Human Nutrition, College of Medicine, Veterinary and Life Science, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study will published in scientific journal upon finished